CLINICAL TRIAL: NCT06632275
Title: Family Caregiver Participation in Hospital Care in a Tertiary Hospital in Bangladesh: a Mixed Methods Study
Brief Title: Family Participation in Bangladesh Hospital Care
Status: Completed | Type: Observational
Sponsor: Michele van Vugt (Other)
Collaborators: Chattogram Medical College Hospital (Unknown); Asian University for Women (Unknown); Mahidol Oxford Tropical Medicine Research Unit (Other); Amsterdam UMC, location AMC (Other)
Responsible Party: Sponsor-Investigator, Michele van Vugt, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: FPBDMM
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Hospitalized Patients
Keywords: Family caregivers; Hospital; Adult; Bangladesh; Family; Care; Mixed method; Observational; Cohort; Prospective; Qualitative; Time and Motion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prospective Observational Cohort: Patient and family caregiver dyads will be recruited for a prospective cohort observation for at least 24 hours and a maximum of seven days. At inclusion, baseline and self-reported data from admission until inclusion will be collected. After inclusion, data will be collected every 24 hours on self-reported outcomes of the last 24 hours. Patients and family caregiver dyads will be followed until discharge, transfer to another department, death or a maximum of seven days of follow-up. If dyads stay longer than seven days, daily follow-up is ended and they are called once 14 days later to collect outcome data.
- Time and Motion: Nurses and doctors will be recruited for time-and-motion observations by a trained non-participant observer during their shift on the medicine ward. Observers will use a REDCap to record where, what, for how long and how health workers perform tasks and interactions during their shifts. Observations will take place in sets of two hours each. Approximate equal amounts of observations will be done on all medicine wards. Observations will occur on different days of the week, at different shifts during the day, and at different times during a shift to collect data from different care contexts. Baseline data of the shift is recorded at the start of the observation.
- Qualitative: The qualitative arm of the study involves interviews and focus group discussions with patients, family caregivers, nurses, doctors and hospital administrators. The FGDs and interviews will be performed in Bengali by a local researcher experienced in qualitative research. An interview guide is used to define themes for the conversations, however, the interviewer is encouraged to follow the flow of the conversation by changing the order of topics or asking additional questions. The main themes of the interview guide are (1) the role of family participation in hospital care, (2) the perceived effect of family participation, (3) the barriers and facilitators for family participation in hospital care, and (4) the opportunities for improving family caregiver participation in hospital care.

SUMMARY:
This mixed methods study aims to understand family care participation in the adult medicine wards of Chattogram Medical College Hospital, Bangladesh. The main questions it aims to answer, from the perspective of the patient, family caregiver, nurse, doctor, ward assistant, and hospital administrator, are:

1. What is the role of the family caregiver in hospital care?
2. What is the perceived effect of family participation in hospital care?
3. What are the barriers and facilitators experienced in family participation?
4. What are suggestions for family participation interventions?

These questions will be answered with three study arms:

1. A prospective observational cohort (population: patients and family caregivers)
2. A time and motion study (population: nurses and doctors)
3. Interviews and focus group discussions (population: patients, family caregivers, nurses, doctors, ward assistants, and hospital administrators)

ELIGIBILITY:
Prospective Observational Cohort

* Inclusion Criteria

  * Population
  * Patient: Admitted to the ward (in-patient)
  * Family caregiver: caregiver providing care at the bedside of the patient on the ward
  * Environment: Admitted to medicine wards 13, 14 or 16 of Chattogram Medical College Hospital
  * Admission time: Admitted in the last 48 hours
  * Adult: ≥18 years
* Exclusion criteria

  * Admission time: Planned discharge or transfer within the first 24 hours of admission
  * Child: <18 years
  * Previously enrolled in this study arm
  * No consent given

Time and Motion

* Inclusion Criteria

  * Population: Nurses and doctors
  * Environment: Working in the medicine wards 13, 14 or 16 of Chattogram Medical College Hospital
* Exclusion Criteria

  * Population: <6 months work experience on wards 13, 14 or 16 of CMCH
  * Previously enrolled in this study arm
  * No consent given

Qualitative (interviews and focus group discussions)

* Inclusion Criteria

  * Population
  * Patient: Admitted to the ward (in-patient)
  * Family caregiver: Caregiver providing care at the bedside of the patient on the ward
  * Health workers: Nurses, doctors and ward assistants
  * Hospital administrator: Managers and professors
  * Environment
  * Patient: Admitted to medicine wards 13, 14 or 16 of CMCH
  * Family caregiver: Caring for their relative on wards 13, 14 or 16 of CMCH
  * Health worker: Working on wards 13, 14 or 16 of CMCH
  * Hospital administrator: Responsible for care delivery on wards 13, 14 or 16 of CMCH
* Exclusion Criteria

  * Population
  * Patient: Unconscious or unable to participate in a conversation
  * Family caregiver: Unable to leave the patient for reasons of safety
  * Health worker: <6 months of work experience on wards 13, 14 or 16 of CMCH
  * Hospital administrator: <6 months in a management role for wards 13, 14 or 16 of CMCH
  * Admission time
  * Patient: Admitted <48 hours
  * Family caregiver: <8 cumulative hours present at patient bedside in last 48 hours
  * Child: <18 years
  * Previously enrolled in this study arm
  * No consent given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes the patients, family caregivers, nurses, doctors, ward assistants, and hospital administrators admitted/caring/working on the general medicine wards of Chattogram Medical College Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 353 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
The role of family participation in hospital care | During admission to the general medicine ward
  The role of family participation will be described with data from:
  1. Prospective observational cohort: patient baseline characteristics, family caregiver baseline characteristics, care characteristics during follow-up (for example: tasks performed, number of caregivers present, hours caregiver is present), end of follow-up status (example: discharged, transferred, death).
  2. Interviews and FDG: with patients, family caregivers, nurses, doctors, ward assistants, and hospital administrators.
The perceived effect of family participation in hospital care | During admission to the general medicine ward
  The perceived effect of family participation will be described with data from:
  1. Time and motion: division of work time of nurses and doctors, time spend interacting with patients and family caregivers.
  2. Interviews and FDG: with patients, family caregivers, nurses, doctors, ward assistants, and hospital administrators.
The barriers and facilitators of family participation in hospital care | During admission to the general medicine ward
  The barriers and facilitators of family participation will be described with data from:
  1. Prospective observational cohort: patient baseline characteristics, family caregiver baseline characteristics, care characteristics during follow-up (for example: tasks performed, number of caregivers present, hours caregiver is present), end of follow-up status (example: discharged, transferred, death).
  2. Time and motion: division of work time of nurses and doctors, time spend interacting with patients and family caregivers.
  3. Interviews and FDG: with patients, family caregivers, nurses, doctors, ward assistants, and hospital administrators.
The intervention suggestions for family participation in hospital care | During admission to the general medicine ward
  The barriers and facilitators of family participation will be described with data from:
  1. Interviews and FDG: with patients, family caregivers, nurses, doctors, ward assistants, and hospital administrators.

CONTACTS AND LOCATIONS:
Locations (1):
- Chattogram Medical College Hospital, Chittagong, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided
Data can be requested from the research group.